CLINICAL TRIAL: NCT05201989
Title: Biomarkers and Epigenetic Markers Associated With Pain in Patients With Symptomatic Atrial Fibrillation Compared With Controls
Brief Title: Biomarkers and Epigenetic Markers Associated With Pain in Patients With Symptomatic Atrial Fibrillation
Acronym: PAIN
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Anna Björkenheim, Principal investigator, Region Örebro County
Other Study IDs: 276727
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Symptoms; Quality of life; Pain
MeSH Terms: conditions — Atrial Fibrillation; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial fibrillation: Subjects with symptomatic paroxysmal atrial fibrillation scheduled for AF ablation at Örebro University hospital
- Control: Sex and age-matched subjects without AF

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia and the number of patients with AF is expected to increase substantially in the coming decades. One third of patients with AF report no AF-associated symptoms, but up to one-fourth report severe symptoms. It is unclear why patients' experience of AF-related symptoms varies so much. We have previously shown that patients with symptomatic AF exhibit lower pain tolerance than patients with asymptomatic AF, as well as impaired pain inhibitory control and facilitated summation of pain, indicating that pain sensitisation may be of importance in symptomatic AF. In patients with chronic pain conditions, several biomarkers and epigenetic markers associated with generation and /or maintenance of chronic pain have been identified. Previous research of biomarkers and epigenetic markers associated with pain is sparse in patients with AF.

The objective is to study levels of biomarkers and epigenetic markers in blood in patients with symptomatic paroxysmal AF (n=100), in relation to severity of AF symptoms, and compared to age- and sex-matched controls without AF (n=100). Blood will be obtained before and after AF ablation and levels of biomarkers, epigenetic markers and cardiac and inflammatory markers, analysed. Patients will complete an AF-specific symptom and a generic health-related quality of life questionnaire.

In the future, biomarkers and epigenetic markers associated with pain may be used as a tool for evaluation of patients with AF and have an impact on individualized management. Another possibility is a rationale for future studies of novel analgesics that neutralize biomarkers or antagonizes its receptors.

ELIGIBILITY:
Inclusion Criteria:

* On waiting list for AF ablation (only symptomatic subjects are offered ablation)
* Paroxysmal AF and persistent AF (AF that is continuously sustained beyond 7 days, including episodes terminated by cardioversion after ≥7 days)
* Written informed consent

Exclusion Criteria:

* Previous pulmonary vein isolation
* Cognitive or psychiatric condition
* Diabetes mellitus
* Ischemic heart disease
* Heart failure
* Asthma
* Pregnancy
* Previous/current drug or alcohol abuse
* Previous neurological or concomitant musculoskeletal disorders
* Continuous analgesic medication

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects who are planned for an AF ablation at Oerebro University Hospital, will be offered the chance to participate in the study. The subjects choice of whether they participate or not will not affect their planned ablation. The waiting list for AF ablation consists of subjects suffering from symptoms due to AF where ablation has been shown to reduce symptoms and improve quality of life.
  100 controls without AF will be recruited through poster advertisements primarily at Oerebro University Hospital, Sweden. If needed, advertisements will be expanded to members of the general public who meet the inclusion criteria in the city of Oerebro, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Biomarkers and epigenetic markers associated with pain | 3 days
  Blood tests will be obtained from subjects the day before, and the day after a planned AF ablation. A total of 30 ml of blood will be obtained at each occasion. The samples will be studied for the association of biomarkers and epigenetic markers to the severity of AF symptoms. Blood samples will be obtained from participants without AF (controls). Biomarkers and epigenetic markers will be compared between the control group and the group with symptomatic AF.

SECONDARY OUTCOMES:
Correlation of age, sex, AF duration, health-related quality of life to biomarkers and epigenetic markers. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Anna Björkenheim, MD, PhD, Principal Investigator — Department of Cardiology, Örebro University Hospital and Örebro University
Locations (1):
- Department of cardiology, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan was shared with Dennis Boye Larsen and Lars Arendt Nielsen in Aalborg, Denmark over e-mail in August 2021. The clinical study report and encoded data regarding patient characteristics and results from questionnaires and blood tests will be shared with Dennis Boye Larsen and Lars Arendt Nielsen in Aalborg, Denmark, for statistical analysis. Data will be made available by an encrypted usb flash drive sent by post. There is no other plan to make individual participant data available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The encoded individual participant data will be available for Dennis Boye Larsen and Lars Arendt Nielsen from 1st January 2022 to the end of September 2023.
Access Criteria: Coded data will be available upon reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT05201989/Prot_SAP_000.pdf